CLINICAL TRIAL: NCT03552172
Title: Retrospective Study of Prescribed Physical Activity in Patients With Overactive Bladder Syndrome Monitored Within the Pelvi-perineology Network in Dijon: Evaluation of Prescription Compliance and Impact on Quality of Life
Acronym: HAV-AP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BUCHOT 2017
Record Dates: First submitted 2018-04-27; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-04

CONDITIONS: iOAB= Idiopathic Overactive Bladder
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prescription physical activity
  Interventions: Other: Physical activity
- No prescription for physical activity or suspension
  Interventions: Other: Absence of or suspended physical activity

INTERVENTIONS:
Other: Physical activity — PHYSICAL ACTIVITY: Rhythm of meetings, number of meetings, place of meetings
  Groups: Prescription physical activity
Other: Absence of or suspended physical activity — the brakes responsible for a stop or lack of practice
  Groups: No prescription for physical activity or suspension

SUMMARY:
Overactive bladder (OAB) is a clinical syndrome defined by the International Continence Society (ICS) and the International Urogynecological Association (IUGA) as urinary urgency (sudden and uncontrollable urge to urinate) possibly associated with urinary frequency (urination greater than 8 times per day), nocturia (2 or more urinations per night) or urinary incontinence (UI). In most cases no root cause is found, so it is referred to as idiopathic overactive bladder (iOAB).

The treatment of iOAB is based primarily on hygiene and dietary measures and perineal rehabilitation. If these are insufficient, medical anticholinergic treatment is offered.

Second-line therapies are based on percutaneous neuromodulation of the tibial nerve, neuromodulation of the sacral roots S3 and intra-detrusor injection of botulinum-A toxin.

iOAB has a significant negative impact on patients' quality of life, particularly in cases of associated urinary incontinence. It is at the origin of low self confidence.

A significant proportion of patients with iOAB are not managed or are not satisfied with treatment.

A strong epidemiological correlation between AVH and metabolic syndrome (MS) was demonstrated in a literature review of 119 articles. MS is a clinical-biological syndrome defined by the National Cholesterol Education Program Adut Treatment Panel III (NCEP ATP III). The prevalence of OAB increases with that of obesity but only from a waist circumference of at least 100cm. S. Boudokhane showed in a prospective study of 34 patients with MS defined by the NCEP ATP III criteria that waist circumference, BMI and post prandial glucose were positively correlated with the presence of OAB measured by the PSU score (p<0.05).

Physical activity (PA) is defined as any body movement produced by skeletal muscles resulting in a substantial increase in energy expenditure above rest energy expenditure (WHO). The efficacy of AP on MS has been demonstrated in primary prevention and treatment of MS by the HERITAGE study and the controlled trial established under the Diabetes Prevention Program (DPP). The follow-up was conducted over 3.2 years and showed a significant decrease in the incidence of MS in the PA group by 41% compared to placebo (p<0.001). The action of PA on iOAB has not been directly studied but some studies have shown that PA and pelvic floor muscle strengthening significantly and respectively decrease the number of mixed (p< 0.0001) (14) or urgency (p=0.009) UI episodes. Since March 2017, the prescription of modified PA is possible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age with iOAB
* The presence of iOAB defined as a positive response (yes, several times a week or several times a day) to the question "how many times in the past 4 weeks have you had to rush to the bathroom to urinate because of an urgent need?
* Treatment unsuccessful or insufficient improvement with discomfort related to OAB on EN>5 by 1st or 2nd line treatments (anticholinergic, alpha-blocker, peripheral neuromodulation by urostim)
* Treatment not changed for 3 months or stopped for at least 4 weeks

Exclusion Criteria:

* Patients with pure stress urinary incontinence or predominantly stress mixed incontinence
* Subjects with neurological diseases (multiple sclerosis, Parkinson's...)
* Subjects with acute urinary tract infection
* Subjects with post micturition residue > 150 mL
* Subjects with untreated bladder obstruction
* Subjects with prolapse grade ≥ 3
* Subjects with painful bladder syndrome
* Subjects who received chemotherapy or radiation therapy
* Subjects conducting self-surveys
* Subjects with cardiovascular factors whose exercise training is not authorized by the cardiologist
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with idiopathic overactive bladder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
ryhthm of physical activity sessions | 3 months
Number of physical activity sessions | 3 months
Location of sessions | 3 months
Quality of life score | Change from basline quality of life at 3 months
Evolution of Discomfort related to urinary disorder | Change from baseline discomfort related to urinary disorder at 3 months
Number of urinations per 24 hours | Change from baseline number of urinations per 24 hours at 3 months
Number of incontinence episodes per 24 hours | Change from baseline number of incontinence episodes per 24 hours at 3 months
OAB Sub-scores on the PSU questionnaire | Change from baseline OAB Sub-scores on the PSU questionnaire at 3 months
Drinking habits according to the urination calendar | Change from baseline drinking habits at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France